CLINICAL TRIAL: NCT05081453
Title: Early Identification and Treatment of Developmental Trochlear Femoral Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joaquín Moya-Angeler Pérez-Mateos (Other)
Responsible Party: Sponsor-Investigator, Joaquín Moya-Angeler Pérez-Mateos, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Organization: Hospital Universitario Virgen de la Arrixaca (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUVArrixaca
Record Dates: First submitted 2021-09-15; First posted 2021-10-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: TROCLEAR DYSPLASIA

STUDY DESIGN:
Intervention Model Description: Parallel controlled triple-blind randomized clinical trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pavlik harness treatment group (Experimental): Application of a pavlik harness for 2 months in position seeking 90º of flexion of both knees and 45º of hip flexion with some abduction. An ultrasound control is performed at 2 and 6 months
  Interventions: Device: pavlik harness
- Control group without intervention (No Intervention): Control group without intervention. An ultrasound control is performed at 2 and 6 months

INTERVENTIONS:
Device: pavlik harness — The application of a pavlik harness will be carried out in the intervention group. It will follow a protocol similar to that of the treatment of hip dysplasia in terms of follow-up and safety
  Arms: Pavlik harness treatment group

SUMMARY:
Title

Early identification and treatment of developmental trochlear femoral dysplasia.

Objectives

To identify developmental trochlear femoral dysplasia (DTFD) in the newborn early after birth by ultrasound and evaluate the effect of its treatment with a modificed Pavlik harness.

Study design

Randomized triple-blind clinical trial.

Study population

Newborns with risk factors for the development of DTFD.

Treatment of subjects

Treatment using a modified Pavlik harness currently used for the treatment of developmental dysplasia of the hip (CDD) over a period of two months.

Variables analyzed

Trochlear groove angles measured by ultrasound before and after the intervention in the treatment group and control group.

Follow-up

Two weeks, eight weeks and six months.

Statistic analysis

Student's t test will be used for related samples to compare and analyze the results of each group at the beginning and after the treatment (intervention group) or follow-up (control group). Study will be triple blinded.

DETAILED DESCRIPTION:
Joint dysplasias consist of alterations in the normal development of a joint. In these cases, the formation of the normally congruent joint surfaces is altered, producing functional abnormalities that, depending on the degree of dysplasia, can lead to a spectrum of clinical manifestations ranging from complete dislocation, subluxations, severe instabilities, and ultimately early osteoarthritis.

The most studied joint dysplasia is developmental dysplasia of the hip (CDD) where the head of the femur and the acetabulum present different degrees of malformation, giving rise to a non-congruent joint. The clinical spectrum of manifestations of this pathology varies from a complete dislocation to milder forms of dysplasia that can manifest in childhood, youth or adulthood as early osteoarthritis, sometimes requiring multiple interventions for its treatment.

Early detection methods for CDD include: the identification of prenatal risk factors (intrauterine position, family history, first-born…), exploration through specific maneuvers, and confirmation by imaging tests such as ultrasound at birth. The early treatment of CDD consists of the application of a Pavlik harness whose purpose is to keep the newborn in a full-time position (frog position) in which the head of the femur remains completely congruent with the acetabulum, allowing the dysplasia to be reversed in early ages. Thanks to these early detection methods and its early treatment (with minimal adverse effects), many of these clinical alterations that previously went unnoticed have been prevented, and whose late treatment involves surgeries with a degree of invasiveness inversely related to the time of detection of DDC.

The knee is another joint susceptible to developing dysplasia. The most frequent dysplasia of the knee joint involves the femoropatellar joint (FP) formed by the patella and the femoral trochlea. Its normal function is vital to be able to flex and extend the leg since the patella acts as a lever arm increasing the strength of the quadriceps. Therefore, it is a joint subjected to high tensile forces.

In the normal knee in extension, the concave patella is located in the most proximal part of the femur without having any contact with the convex femoral trochlea. As the knee is bent, the patella runs into the deep femoral groove (normal groove angle 135º), which acts as containment and allows it to slide distally as the knee is bent further. It is in these knee flexion positions, more than 90º, where there exist more tensional forces between both articular surfaces.

Developmental trochlear femoral dysplasia (DTFD), therefore, consists of the abnormal development of both articular surfaces resulting in a non-congruent joint. However, unlike CDD, it is not detected early since it generally manifests in adolescence in the form of recurrent dislocations with minimal trauma in severe cases. Recurrent patellar dislocations are a serious and complex problem for both the patient and the surgeon since in adolescence it is not possible to reverse DTFD and surgeries to generate a normal trochlear groove (trochleoplasty) can have catastrophic results generating disability and lameness for life in a not inconsiderable percentage of patients. Milder forms of dysplasia that do not appear in adolescence produce instabilities or subluxations and alterations in the patellar tracking that trigger recurrent knee pain and often end up producing early osteoarthritis in young patients. The treatment of this type of patient is also not very rewarding and sometimes they require surgeries at an early age with poor results.

The fact that DTFD manifests itself late during adolescence, has biased the scientific community to focus its efforts on research related to the surgical treatment of this pathology and not on its prevention at an early age, as is the case with DDC. However, more recent studies are focusing their objectives on the early detection and etiological analysis of this structural anomaly in order to prevent it. Specifically, investigators conducted a study in newborns with early ultrasound in order to identify risk factors related to PRDD. These investigators concluded that the intrauterine breech position at birth was 45 times more likely to develop DTFD than the cephalic position.

Although the etiology of DTFD is not clear, more and more studies point to the idea that the lack of a mechanical stimulus by the patella in the femoral sulcus causes both articular surfaces not to develop normally. According to a study that developed an experimental study in newborn rats resecting the patella, the morphological development of the femoral trochlea is influenced by its abnormal mechanical stress. This hypothesis has also been reinforced by the work of other investigators where, in an experimental study in growing rabbits, they observed the development of DTFD in those rabbits in which they produced a permanent patella dislocation (avoiding the contact of the patella on the femoral trochlea). These findings would also justify those previously described by where it was observed that those newborns in a breech position with their legs extended (in extension, the patella is located proximal to the femoral groove and does not exert the mechanical stimulus necessary for normal groove development) had a higher incidence of DTFD.

These investigations support the hypothesis that the absence of mechanical stimulation of the patella on the femoral trochlea leads to an alteration in its development, producing DTFD. This situation led two different researchers to carry out different studies in order to find out whether in those cases with DTFD, dysplasia could be reversed by returning the mechanical stimulus of the patella to the trochlea. A study demonstrated that dislocation and subsequent reduction of the patellofemoral joint could reverse DTFD in growing rabbits and other investigators showed that realignment surgery could remodel the dysplastic trochlea at very young ages in a human clinical study after an eleven-year follow-up.

These findings suggest that it is possible to identify DTFD early in newborns with risk factors using ultrasound and that there is the possibility of modeling the dysplastic trochlea if the necessary mechanical stimulation is achieved by the patella. However, although there is evidence that this situation can be reversed, so far no clinical study has been developed in neonates with DTFD to assess the effect of different interventions. Currently, it is more than known that keeping the knee at 90º of flexion is when there are greater contact forces between the patella and the trochlea. As in DDC, this position could be maintained in newborns with DTFD by using a harness, with the intention of achieving constant and permanent mechanical stimulation of the patella on the dysplastic trochlea that allows modeling the dysplastic groove. during the early growth phase.

That is why the investigators propose the development of a randomized, double-blind clinical trial with the aim of early identification by ultrasound of newborns with risk factors for the development of DTFD and subsequently evaluate the result of treatment with a harness that maintains the knee at 90º flexion for two months.

The hypothesis under study is based on the fact that early identification and treatment of DTFD in newborns using a harness could model the dysplastic trochlea and prevent this malformation and its consequences in the short and long term, as is the case with DDC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term and preterm newborns > 35 weeks
* Breech presentation at birth.

Exclusion Criteria:

* Infant cerebral palsy,
* Developmental disorders
* Chromosomal diseases.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
measurement of the angle of the trochlear groove | 20 minutes
  It is performed with ultrasound on the subject's knee. It is carried out by orienting the axis of the leg with the transverse probe. The image is focused on the ossified nucleus of the distal femur and oriented so that both non-ossified femoral condyles are visible. The measurement of the angle of the trochlear groove is taken from the nadir of the trochlea along the lines of best fit of the medial and lateral walls of the trochlea.

SECONDARY OUTCOMES:
patellar height | 15 minutes
  It is performed by orienting the ultrasound probe in the sagittal plane to obtain measurements of the patella and patellar tendon

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Publication of the study results in journals related to the specific topic

REFERENCES:
- [Result] Gray CJ, Shanahan MM. Breech Presentation. 2022 Nov 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448063/ PMID 28846227
- [Result] Oye CR, Foss OA, Holen KJ. Breech presentation is a risk factor for dysplasia of the femoral trochlea. Acta Orthop. 2016 Feb;87(1):17-21. doi: 10.3109/17453674.2015.1089023. Epub 2015 Sep 18. PMID 26381593
- [Result] Oye CR, Foss OA, Holen KJ. Minor change in the sulcus angle during the first six years of life: a prospective study of the femoral trochlea development in dysplastic and normal knees. J Child Orthop. 2018 Jun 1;12(3):245-250. doi: 10.1302/1863-2548.12.180026. PMID 29951124
- [Result] Onor GI Jr, Yalcin S, Kaar SG, Pace JL, Ferrua P, Farrow LD. The Evaluation of Trochlear Osseous Morphology: An Epidemiologic Study. Orthop J Sports Med. 2021 Apr 2;9(4):2325967121994548. doi: 10.1177/2325967121994548. eCollection 2021 Apr. PMID 33869646